CLINICAL TRIAL: NCT00004861
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of CI-994 Capsules Plus Gemcitabine Infusion Versus Placebo Capsules Plus Gemcitabine Infusion in the Treatment of Patients With Advanced Pancreatic Cancer
Brief Title: Gemcitabine With or Without CI-994 in Treating Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: PD-994-011; CDR0000067513; ILEX-994-011
Record Dates: First submitted 2000-03-07; First posted 2004-06-18 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas; stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; tacedinaline

INTERVENTIONS:
Drug: gemcitabine hydrochloride
Drug: tacedinaline

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug or giving drugs in different ways may kill more tumor cells.

PURPOSE: Randomized phase II trial to compare the effectiveness of gemcitabine with or without CI-994 in treating patients who have advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the efficacy and safety of CI-994 given in combination with gemcitabine compared to gemcitabine alone in the treatment of patients with advanced pancreatic cancer.

OUTLINE: Gemcitabine is the standard of care for pancreatic cancer and is administered by intravenous injection. Patients receive gemcitabine once a week for 3 weeks followed by 1 week of rest. Patients take the capsules (placebo or investigational chemotherapy) daily for 21 consecutive days beginning with the first gemcitabine infusion. The duration of treatment is determined by the patient's tolerance of therapy and the assessment of disease response.

PROJECTED ACCRUAL: A total of 172 patients will be enrolled in Canada, Europe, and the United States on a competitive basis.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologic or cytologic diagnosis of advanced (stage II or III) or metastatic (stage IV) adenocarcinoma of the exocrine pancreas and not considered a surgical candidate Measurable or unmeasurable disease

PATIENT CHARACTERISTICS: Age: Age greater than or equal to 18 years Performance status: Karnofsky 70-100% Life expectancy: Expected survival greater than 12 weeks Hematopoietic: No inadequate bone marrow function within 2 weeks prior to randomization as evidenced by the following: Absolute neutrophil count less than 2000/mm3 Platelet count less than 100,000/mm3 Hepatic: No inadequate hepatic function within 2 weeks prior to randomization as evidenced by the following: Total bilirubin greater than 1.5 times upper limit of normal (ULN) AST or ALT greater than 3 times ULN (greater than 5 times ULN if liver metastases is documented) Renal: No inadequate renal function within 2 weeks prior to randomization as evidenced by the following: Creatinine clearance less than 50 mL/min Other: Adequate IV access to receive gemcitabine infusion Capable of swallowing intact study medication capsules Capable of giving informed consent Capable of following instructions or having a daily caregiver who assumes responsibility for administering study medication and completing medication diaries No life threatening illness (unrelated to tumor) No women of childbearing potential unless using an acceptable method of contraception, or who are pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior immunotherapy or biologic therapy may be allowed, but must have been completed at least 1 month prior to randomization Chemotherapy: No prior chemotherapy for advanced stage pancreatic cancer Fluorouracil (with or without leucovorin calcium or interferon) given with radiation as a radiation sensitizer may be allowed, but must have been completed at least 3 months prior to randomization Endocrine therapy: Prior hormonal therapy may be allowed, but must have been completed at least 1 month prior to randomization Radiotherapy: No radiation therapy within 4 weeks prior to first treatment Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-10; Study Completion 2001-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathy M. Diener, PharmD, Study Chair — Pfizer Incorporated - Ann Arbor
Locations (16):
- United States (11):
  - Cedars-Sinai Comprehensive Cancer Center, Los Angeles, California
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - Raleigh Hematology/Oncology Associates - Wake Practice, Raleigh, North Carolina
  - Jewish Hospital of Cincinnati, Inc., Cincinnati, Ohio
  - Ireland Cancer Center, Cleveland, Ohio
  - West Clinic, P.C., Memphis, Tennessee
  - Sarah Cannon-Minnie Pearl Cancer Center, Nashville, Tennessee
  - Tyler Cancer Center, Tyler, Texas
  - Northern Virginia Oncology Group, Fairfax, Virginia
- Canada (5):
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Ottawa Regional Cancer Center - General Division, Ottawa, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec